CLINICAL TRIAL: NCT01066013
Title: Antimicrobial De-escalation Strategy in Medical Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fraser Health (Other)
Collaborators: Vancouver Foundation (Other)
Responsible Party: Anisha Lakhani, Fraser Health Authority
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FHREB 2009-093
Record Dates: First submitted 2010-02-01; First posted 2010-02-10 (Estimated); Last update posted 2010-08-18 (Estimated); Status verified 2010-01

CONDITIONS: Infections
Keywords: Antimicrobial De escalation; Meropenem; Piperacillin tazobactam; Medical patients; Appropriate use; Cost savings; Antimicrobial De-escalation strategy
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prospective Antimicrobial de-escalation arm (Experimental): Antimicrobial de escalation team will assess therapy and make recommendations to (a) change to antibiotic(s) with narrow spectrum,(b) stop antibiotics, (c) order new cultures/investigations or (d) consult with specialists or ID service for full evaluation (if patient's condition is worsening).
  Interventions: Other: Antimicrobial de-escalation strategy
- Restrospective control arm (No Intervention): The control subjects will be drawn from historic data of patients on the same medical unit(s) and will be matched based on age, antibiotics, sex, and infectious diseases diagnosis.

INTERVENTIONS:
Other: Antimicrobial de-escalation strategy — The antimicrobial de-escalation team will record recommendations for de-escalation in the patient's progress notes for the attending physicians to review and act upon as appropriate. The attending physician will be responsible for making changes to antimicrobial therapy and following up on patient progress as per the usual practice.
  Arms: Prospective Antimicrobial de-escalation arm

SUMMARY:
The purpose of this pilot study is to assess the impact of an antibiotic de-escalation strategy on the clinical outcomes (clinical cure or improvement) of medical patients related to the usage of of broad-spectrum antimicrobial agents.

DETAILED DESCRIPTION:
This is an open-label, case-control, pilot study involving medical patients with serious infections who are prescribed meropenem or piperacillin/tazobactam, at Surrey Memorial Hospital. Patients in the experimental arm (cases) will be required to provide an informed consent. A team consisting of an infectious diseases specialist, medical microbiologist and clinical pharmacists will prospectively assess antimicrobial therapy in the enrolled subjects in the prospective arm and make recommendations for antimicrobial de-escalation.

The control group will consist of subjects drawn from historic data of patients on the same medical unit(s) who will be matched based on age, sex, use of broadspectrum antibiotics (meropenem or piperacillin/tazobactam) and infectious diseases diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years and over
* Suspected or confirmed infection for which a Meropenem and/or Piperacillin/Tazobactam is prescribed. This will include any patient who is other concomitant antibiotic(s) such as Vancomycin
* Subject admitted to SMH medical unit(s)
* Pregnant patient (or patients wishing to become pregnant)

Exclusion Criteria:

* Age less than 19 years
* Granulocytopenia (< 1x109/L)
* Allergy or intolerance to meropenem or piperacillin-tazobactam.
* Febrile Neutropenia
* Cystic Fibrosis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-05 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients who had therapy with meropenem or piperacillin/tazobactam de-escalated by the de-escalation team. | 7 days

SECONDARY OUTCOMES:
Clinical efficacy (clinical improvement or complete resolution of infection) | 7 days
Appropriateness of broadspectrum antibiotic (meropenem or piperacillin/tazobactam) prior to de-escalation | 7 days
Cost and consumption (usage data) of antibiotics | 7 days
All cause mortality | 14 days
Length of stay in the hospital | 14 days